CLINICAL TRIAL: NCT02314832
Title: Comparison Between the Risk Falls After Total Knee Arthroplasty With Use of Femoral Nerve Block Versus Adductor Canal Block
Brief Title: Risk of Falling After CFNB Versus ACB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 820115
Record Dates: First submitted 2014-07-01; First posted 2014-12-11 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Falls; Total Knee Arthroplasty (TKA); Osteoarthritis
Keywords: femoral nerve block; adductor canal block; tinetti score; 2- Results to time to up and go (TUG ) test; 3- Results to Tinetti test; 4- Ambulation distance; 5- Pain scores at rest and with movement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous femoral nerve block (Active Comparator): patients receiving continuous femoral nerve block for analgesia after total knee arthroplasty
  Interventions: Procedure: femoral nerve block
- adductor canal block (Active Comparator): adductor canal block group will receive adductor canal block for analgesia after TKA
  Interventions: Procedure: adductor canal block

INTERVENTIONS:
Procedure: adductor canal block — ultrasound guided saphenous nerve block in the adductor canal
  Arms: adductor canal block
Procedure: femoral nerve block — ultrasound guided femoral nerve block
  Arms: Continuous femoral nerve block

SUMMARY:
Blocking sensation from the femoral nerve by injecting local anesthetic around the nerve plays an important role in pain control after total knee replacement. However, femoral nerve block has been associated with increased risk of falls due to weakness of the thigh muscle. This prospective, randomized controlled trial asks the question whether blocking the more distal branch of the femoral nerve (saphenous nerve) will result in less muscle motor block, and thus less risk of falls. The study also aims to compare pain control after both techniques.

DETAILED DESCRIPTION:
If the patient is willing to participate and signs the consent, he/she will be randomized to one of the two treatment groups:

1. Femoral nerve block
2. Adductor canal block

The standard of care anesthesia regimen for this surgery is as follows:

All Patients will receive their Multimodal Perioperative Pain Protocol (MP3) medication as per routine care in the patient receiving area. All blocks are performed in the pre-operative holding area with standard ASA monitors applied. Typically, patients receive 1-2 mg of midazolam and 50-100 mcg of fentanyl for sedation during the placement of the block. Standard operating procedure of the block room will be followed. Block time out will be preformed according to standard operating procedure. All blocks will be done under ultrasound guidance. Sonosite (S nerve) machine will be used with a high frequency linear (HFL) US probe with 6-13 MHZ frequency. Both CFNB and ACB will take be performed according to the SOP in the investigators department.

For CFNB: Images of the femoral nerve will be obtained in the short axis. 1% lidocaine will be used for local infiltration of the skin. A 2 inch 18 G touhy needle ( B Braun) will be advanced in plane under US guidance . Confirmation may take place with Quadricpes muscle twitches and patella movement between 0.3 and 0.4mA (2Hz; 0.1ms). A bolus of 20 ml of Ropivicaine 0.5% will be injected. A non stimulating catheter will be advanced through the needle to a distance of 3-4 cm beyond the needle tip. Catheter will be secured in place using benzoin, Steristrips, and a tegaderm.

For the ACB: ultrasound survey at the medial part of the thigh will take place, halfway between the superior anterior iliac spine and the patella. In a short axis view, the femoral artery will be identified underneath the sartorius muscle, with the vein just inferior and the saphenous nerve just lateral to the artery. The needle will be introduced in-plane and 2 to 3 mL of LA bolus (0.2% ropivicaine) will be used to verify correct placement of the needle in the vicinity of the saphenous nerve in the adductor canal. A bolus of total volume of 20 ml of Ropivicaine 0.5% will be injected through the needle. The catheter will then be introduced and advanced 2-3 cm beyond the tip of the needle.

At the conclusion of surgery a large obaque dressing will be applied from the femoral crease to the mid thigh region so that the catheter location will be concealed. Both catheters will be connected to a pump that will infuse local anesthetic. Ropivicaine 0.2% at 8 ml/hour. There is usually a period of time before the patient transport to the operating room during which the investigators will be able to evaluate if the block is effective and sufficient for surgery.

Patients will receive either general or spinal anesthesia in the operating room. All patients will receive prophylaxis for nausea and vomiting during surgery. Regimen for prophylaxis include a single dose of dexamethasone after induction of anesthesia and a single dose of Ondansetron 20 minutes before recovery from anesthesia. This study is not deviating from the standard of care anesthetic regimen for this surgical procedure at Penn Presbyterian Medical Center. Only the type of blocks will be different between the two groups.

Postoperative analgesia All PACU analgesia will follow standard of care protocol for post operative care at PPMC. Hydromorphone 0.2 mg iv q5 minutes as necessary. The infusion of the local anesthetic will start in the PACU.

In the PACU, patients are assessed for pain with the Visual Analog Scale (pain scale of 1 to 10) at routine time points for the duration of their stay. The worse VAS score will be recorded.

Postoperative Analgesia

Postoperative analgesia will follow the MP3 protocol. The protocol includes administration of around the clock acetaminophen, Celebrex, gabapentin, immediate and extended release oxycodone.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for primary total knee arthroplasty
* American Society of Anesthesiologists (ASA) physical status I -III
* mentally competent and able to give consent for enrollment in the study

Exclusion Criteria:

1. Patient younger than 18 years old
2. Allergy to local anesthetics, systemic opioids (fentanyl, morphine, hydromorphone, and any of the drugs included in the multimodal perioperative pain protocol (MP3).
3. Revision surgery will be excluded.
4. Impaired kidney functions and patient with coagulopathy will also be excluded.
5. Chronic pain syndromes; Patients will be defined to have chronic pain if they are using regular daily doses of systemic narcotics for the past 3 months prior to the surgery.
6. BMI of 40 or more
7. Pregnancy (positive urine pregnancy test result in Preop area on morning of surgery)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
risk of falling score | 24 hours after surgery
  The percentage of patients at high risk of falls as evaluated by Tinetti score in both groups.
  Scores of 19 or less are usually associated with higher risk of falls.

SECONDARY OUTCOMES:
Pain scores | 48 hours
  pain scores at rest and with movement

CONTACTS AND LOCATIONS:
Overall Officials: Nabil M Elkassabany, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States